CLINICAL TRIAL: NCT03640026
Title: Glucose Disorders Induced by Tacrolimus on Pre Transplantation Endstage Renal Disease Patients
Acronym: GLITTER
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Centre Hospitalier Departemental Vendee (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CHD045-17
Record Dates: First submitted 2018-08-17; First posted 2018-08-21 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-04

CONDITIONS: Kidney Failure, Chronic
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Tacrolimus treatment (Experimental)
  Interventions: Drug: Tacrolimus

INTERVENTIONS:
Drug: Tacrolimus — Tacrolimus will be initiated at 0.1 mg/kg/day in two separate 12-hour oral doses (capsules) for 14 days.

SUMMARY:
Diabetes after kidney transplantation is a frequent complication, the incidence of which varies from 7 to 45% depending on the studies and on the diagnostic criteria used. Post-transplant diabetes is an early complication, most often occurring in the first month after transplantation.

In addition to the additional health costs generated by the appearance of post-transplant diabetes, the risk of graft loss is increased by 60% and the overall mortality risk by 90%. Similarly, the development of glucose intolerance after transplantation is associated with higher mortality.

Tacrolimus treatment is therefore currently one of the most important risk factors for diabetes at the time of transplantation.

Indeed, several in vitro and in vivo animal studies have shown that tacrolimus alters pancreatic endocrine function.

In the final stage, this cellular toxicity leads to diabetes, most often diagnosed on the rise in capillary or venous blood sugar levels after transplantation. This diabetes often requires hypoglycemic treatment with insulin or oral anti-diabetic drugs. for a variable period. The pro-diabetogenic effect of tacrolimus is sometimes irreversible, justifying preventive treatment.

No clinical studies have looked at "sub-clinical" changes in insulin secretion or insulin resistance under tacrolimus prior to the onset of diabetes. The static indices HOMA-β% and HOMA-IR (Homeostasis Model Accessment of insulin resistance) make it possible to estimate insulin secretion and insulin resistance in fasting patients respectively, while the oral glucose disposition index (IDO) makes it possible to study insulin secretion and action dynamically (after a 75 g glucose load), and are calculated as follows:

HOMA IR= Fasting blood glucose (mmol/L) x Fasting insulin (mU/L)/ 22.5 HOMAβ% = 20 x fasting insulinemia (mU/L) / fasting plasma glucose (mmol/L) - 3.5 IDO = (delta insulinemia T30-T0/ delta blood glucose T30-T0)/insulinemia T0

These indices have already been studied in dialysis patients (diabetic and non-diabetic) and may allow a more detailed study of pancreatic response and insulin resistance under tacrolimus in patients prior to renal transplantation. Determining the "pancreatic response" to tacrolimus in patients prior to transplantation would prevent diabetes by adapting immunosuppressive treatment and post-transplant screening modalities in the event of pre-transplant subclinical abnormalities identified in our study. The development of tacrolimus-induced diabetes in pre-transplantation in our study will be a contraindication to tacrolimus at the time of transplantation and ciclosporin therapy will be preferred.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patient eligible for kidney transplantation at the Nantes University Hospital
* Hemodialysis patient in one of the participating centres
* Patient who is able to understand the proposed protocol and has given free and informed consent
* Patient with affiliation to the French social security system.

Exclusion Criteria:

* Personal history of diabetes treated or untreated
* Temporary contraindication for carcinological reasons
* Immunosuppressive treatment in the 6 months prior to inclusion
* Macrolide Allergies
* Hypersensitivity to the excipients used in the composition of tacrolimus
* Intolerance to the HGPO test
* Progressive infectious outbreak
* Hepatic insufficiency
* Intercurrent infectious pathology
* Patient under guardianship, curatorship, legal protection measure, or deprived of liberty
* Pregnant women, breastfeeding, or non-menopausal woman who refuses contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-03-08 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Proportion of haemodialysis patients modifying their glycemic profile receiving Tacrolimus | During 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Awena LE FUR, Principal Investigator — CHD Vendée
Locations (2):
- France (2):
  - Centre Hospitalier Départemental Vendée, La Roche-sur-Yon
  - Centre Hospitalier Universitaire Nantes, Nantes